CLINICAL TRIAL: NCT06173934
Title: The Effect of Gastric Emptying on Blood Glucose Profile of Type 1 Diabetes Mellitus and Its Therapeutic Strategies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY20230915-11
Record Dates: First submitted 2023-12-06; First posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with rapid gastric emptying (Experimental): Patients with rapid gastric emptying
  Interventions: Drug: insulin injection 15 minutes before meals
- Patients with slow gastric emptying (Experimental): Patients with slow gastric emptying
  Interventions: Drug: Insulin injection 15 minutes after eating

INTERVENTIONS:
Drug: insulin injection 15 minutes before meals — Adjust insulin injection time to observe blood glucose spectrum
  Other Names: insulin regulation
  Arms: Patients with rapid gastric emptying
Drug: Insulin injection 15 minutes after eating — Adjust insulin injection time to observe blood glucose spectrum
  Other Names: insulin regulation
  Arms: Patients with slow gastric emptying

SUMMARY:
Establish a cohort study to describe the characteristics of gastric emptying in patients with type 1 diabetes, and adjust the timing of insulin injection during meals to improve blood glucose fluctuations according to the speed of gastric emptying.

DETAILED DESCRIPTION:
1. T1DM that met the inclusion criteria was tested with baseline blood routine, biochemical and complication screening, and FGM monitoring for 14 days (patient blindness) on the basis of the original regimen (insulin pump or basic insulin combined with fast-acting insulin before three meals); A stable diet should be maintained before and during the study.

1. T1DM that met the inclusion criteria was tested with baseline blood routine, biochemical and complication screening, and FGM monitoring for 14 days (patient blindness) on the basis of the original regimen (insulin pump or basic insulin combined with fast-acting insulin before three meals); A stable diet should be maintained before and during the study.
2. On the 7th day of FGM monitoring, 13C-GEBT examination was performed on an empty stomach;
3. Starting from day 8, patients were divided into groups according to the comparison of gastric emptying T50 with pre-experimental healthy people. Group A, patients with rapid gastric emptying, adjusted the time of fast-acting insulin injection to 15 minutes before meals; Group B, patients with slow gastric emptying, adjusted the time of fast-acting insulin injection to 15 minutes after eating.
4. FGM monitoring was completed on the 14th day and the study was concluded. 2. On the 7th day of FGM monitoring, 13C-GEBT examination was performed on an empty stomach;

3. Starting from day 8, patients were divided into groups according to the comparison of gastric emptying T50 with pre-experimental healthy people. Group A, patients with rapid gastric emptying, adjusted the time of fast-acting insulin injection to 15 minutes before meals; Group B, patients with slow gastric emptying, adjusted the time of fast-acting insulin injection to 15 minutes after eating.

4. FGM monitoring was completed on the 14th day and the study was concluded.

ELIGIBILITY:
Inclusion Criteria:

* 1.Volunteer and sign subject informed consent prior to the trial.

  2.Patients with type 1 diabetes, aged less than 70 years, 7%≤HbA1c≤9.0%.

  3.There were no acute complications such as diabetic ketoacidosis and diabetic hypertonic syndrome.

  4.Subjects were able and willing to undergo 14-day scanning blood glucose monitoring, diet and exercise routine.

Exclusion Criteria:

* 1.Patients with severe gastrointestinal symptoms, history of gastrointestinal disease, surgical history, or impaired liver and kidney function.

  2.Patients who have used drugs that affect gastrointestinal function or appetite in the last week.

  3.History of drug abuse and alcohol dependence within the past 5 years.

  4.Systemic hormone therapy was used in the last three months.

  5.Patients with poor compliance, irregular diet and exercise.

  6.Patients with infection and stress within four weeks.

  7.Patients who could not tolerate 14-day scanning blood glucose monitoring.

  8.Patients who are pregnant, nursing or intending to become pregnant.

  9.Any other obvious condition or comorbidities determined by the investigator: such as serious cardiopulmonary disease, endocrine disease, neurological, neoplastic, other pancreatic disease, history of mental illness.

Max Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Characteristics of gastric emptying(the gastric half-emptying time ) in patients with type 1 diabetes. | 1, 2, 3 years
  Correlation of gastric emptying with disease course, blood glucose fluctuation and complications.

SECONDARY OUTCOMES:
The blood glucose | 1, 2, 3 years
  According to the speed of gastric emptying, the time of insulin injection during meals is adjusted to observe MBG

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Ma, Principal Investigator — Nanjing Medical University affiliated Nanjing First Hospital
Locations (1):
- Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu, China